CLINICAL TRIAL: NCT06098755
Title: Transcendence Research: Holistic Education For Colonized Countries Primarily English Speaking
Brief Title: The Sequestration of Holistic Stress Management Techniques for Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Goddess Zena I. Jones (Other)
Responsible Party: Sponsor-Investigator, Goddess Zena I. Jones, PD/PI, Virtual Tribunal Monastery
Organization: Virtual Tribunal Monastery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RYXWWMJUDPM6
Record Dates: First submitted 2023-10-12; First posted 2023-10-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Stress, Job; PTSD; Hypervigilance; Hyperthyroidism; Migraine; Migraine With Aura; Immunodeficiency; Sickle Cell Trait; Sickle Cell Disease; Anemia, Sickle Cell; Anemia; Fatigue; Anxiety; Depression; Flat Feet; Lordosis; TBI (Traumatic Brain Injury); Rheumatoid Arthritis; Arthritis; Masturbation; Priapism; Erectile Dysfunction; Flight Reaction; Hypertension; Sexual Arousal Disorder; Hemorrhoids; Fibroid
MeSH Terms: conditions — Occupational Stress; Stress Disorders, Post-Traumatic; Hyperthyroidism; Migraine Disorders; Migraine with Aura; Immunologic Deficiency Syndromes; Sickle Cell Trait; Anemia, Sickle Cell; Anemia; Fatigue; Anxiety Disorders; Depression; Flatfoot; Lordosis; Brain Injuries, Traumatic; Arthritis, Rheumatoid; Arthritis; Masturbation; Priapism; Erectile Dysfunction; Escape Reaction; Hypertension; Sexual Dysfunctions, Psychological; Hemorrhoids; Leiomyoma | interventions — Holistic Health

STUDY DESIGN:
Intervention Model Description: Holistic Medicine, also known as Holistic Education, represents a nonclinical approach to healing, recovery and wellness. It focuses on nurturing the whole person-mind, body, and spirit-to achieve optimal well-being. Other names for this intervention include Nonclinical Variables, Transcendence Research and Adult Education.
  The Patient-Centered Medical Home (PCMH) model plays a crucial role in delivering holistic care. PCMH provides individualized care, patient engagement, and comprehensive care coordination within a single practice. The ultimate goal is to improve quality of life through prevention education, treatment, and rehabilitation programs tailored to individual patient needs.
  Holistic Medicine (Holistic Education) emphasizes patient self-help and self-care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resource Utilization Group (Experimental): nonclinical variables
  Interventions: Behavioral: Holistic Medicine (HM)

INTERVENTIONS:
Behavioral: Holistic Medicine (HM) — With informed consent the participant act as a partner to their health and acknowledges responsibility for self-help or self-care directed activities in a non-clinical setting. Transcendence in research involves actively exploring the best possible options or resources for a resolution or self-determination or hypotheses. To reinforce healthy activities, periodic forecast consist of one or more of the following variables: pastoral counseling, lectures, group discussions, sound therapy sessions, team building exercises, faith-based initiatives, outdoor exercise, walking group, support group, supportive care, cooking class, critical thinking questioning and self-assessment tests. Adult content variables are classified under Respite (i.e. adult time, gaming, dance therapy, music therapy, clothing model therapy, civil-branding role-play, interactive Spiritual story) TO (Time-Out).
  Other Names: Holistic Education; Transcendence Research; Adult Education

SUMMARY:
This remote study is intended to assist the population with access to cost-effective pastoral counseling for stress management in the workplace and every day life. Holistic medicine (also known as Holistic Education) doesn't replace nor substitute clinical diagnosis, clinical medical treatment, and clinically prescribed medication. HUMANITARIAN VETERANS ASSOCIATION serves as the tax-exempt peer-review board and Liaison.

DETAILED DESCRIPTION:
The Headmistress or Headmaster is a licensed referral, ordering, and Holistic Medicine prescribing provider only. While a massage chair is considered an expensive preference to reduce stress and for immediate relief; in an economical sense, being able to emotionally adjust to changes and different environments may require self-help practice. With a Holistic approach to wellness, healing and recovery, the 'Whole Person' concept includes biofeedback (i.e. A Pulse MD finger monitor, portable automatic blood pressure monitor, and a contactless infrared thermometer) to document vital signs.

With emphasis on the "Whole Person Concept' mind, body, and spirit, Holistic Medicine (also known as Holistic Education) serves the purpose to provide a holistic approach to healing and recovery through self-help and self-care directed activities. Holistic Medicine is a vital integrative component in today's alternative health care system that doesn't replace nor substitute clinical diagnosis, clinical treatment, and clinically-prescribed medications. Holistic Medicine is a nonclinical Holistic Healthcare option and mostly practiced in Faith-based Initiatives.

The Humanitarian Veterans Association was founded in the year 2011. Over 100 Humanitarian Veterans Association members were recruited in-person at various military/veteran events and support services. Humanitarian Veterans Association Doing Business As Veterans Corps of Humanitarian Veterans Association also serves as the tax-exempt Liaison and Peer-Review Board.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried Couples, Bachelor, and Bachelorette Alaska Medicaid recipients age 22 years old and older.
* Copies of most recent STIs (Sexually-Transmitted Infections) and Drug Panel results
* Must be competent (of sound mind and judgement) and be mobile (physically-active)
* Acknowledge smoke-free, drug-free, and alcohol-free church policy
* Must have access to the Internet, Holy Bible (KJV), and an audio-recorder
* Religious or spiritual belief in prayer meditation for faith-based healing
* Must acknowledge the existence of ethical standards of practice similar to the Hippocratic Oath
* Due to a new tool in the Toolkit: DOGS HELP TO DETECT COVID-19, a negative COVID-19 test may be required at any time whenever COVID-19 is suspected without remedy.

Exclusion Criteria:

* Noncompliance to Inclusion Criteria.
* Married relationship status
* Gender Conversion
* Repeat offenders
* Smokers, vapors, alcoholics, drug abusers.
* Non-Believers in Christian religious practices or prayer.
* Ineligible for Alaska Medicaid
* Immobility
* Diseases without clinical diagnosis, medical treatment, and remedy.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Holistic Medicine Qualitative Method | 1 year
  Qualitative data are not expressed numerically. Qualitative evaluation method summarize evidence from instructed methods of data collection relevant to socioeconomic factors, naturalistic observation, and existing records. Hierarchy scales of evaluation determine client wellness stages and identify areas requiring additional nonclinical variables for optimum wellness.
Holistic Medicine Quantitative Method | 1 year
  Based on an average score total 1-100 point scale questionnaire, self-assessment, and/or critique forms will be used to measure socioeconomic factors as well as behaviors, impact, reaction, coping, etc...

CONTACTS AND LOCATIONS:
Overall Officials: Jones, Study Chair — Humanitarian Veterans Association
Locations (1):
- Virtual Tribunal Monastery, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones G. Transcendence Research: Holistic Healthcare for At-Risk Homelessness Pursuant to Chronic Health Conditions. Transcendence Research. 2025 December; 1(1).
- [Background] Jones G. Transcendence Research: Counterterrorism to Prevent Victimization. Transcendence Research: Holistic Healthcare for At-Risk Homelessness Pursuant to Chronic Health Conditions. 2025 December; 1(2).
- [Result] Jones G. Transcendence Research: Holistic Healthcare for Social-Welfare Inequities Pursuant to Chronic Health Conditions. Transcendence Research: Holistic Healthcare for At-Risk Homelessness Pursuant to Chronic Health Conditions. 2026 January; 2(1).
- See also: Virtual Tribunal Monastery Facility website link — https://virtualtribunalmonastery.vhx.tv/
- See also: DOGS HELP DETECT COVID-19 — https://www.cdcfoundation.org/stories/project-uses-dogs-detect-covid-19
- See also: Dry or Damp Community references — https://www.commerce.alaska.gov/web/amco/AlcoholLocalOption.aspx
- See also: Adult Education — https://en.wikipedia.org/wiki/Adult_education
- See also: Holistic Education (also known as Holistic Medicine) GREEK HIPPOCRATIC OATH — https://www.nlm.nih.gov/hmd/greek/greek_oath.html
- See also: Ecclesiastical Law for the church — https://thelawdictionary.org/ecclesiastical-law/
- See also: MASLOW'S HIERARCHY OF NEEDS PYRAMID e.g.Transcendence Research, Inductive Reasoning (also known as the BOTTOM-UP ANALYSIS) — https://en.wikipedia.org/wiki/Maslow%27s_hierarchy_of_needs
- See also: Self-efficacy — https://en.wikipedia.org/wiki/Self-efficacy
- See also: White House Faith-based & Community Initiative — https://georgewbush-whitehouse.archives.gov/government/fbci/president-initiative.html
- See also: Request for and Consent to Release Information from Individual's Records — https://www.va.gov/find-forms/about-form-3288/
- See also: Consenting Adults Form to Watch Adult Content, Discuss Adult Content, and Participate in Adult Content — https://eforms.com/images/2017/08/Sexual-Consent-Form.pdf
- See also: Means-Tested Benefits — https://studentaid.gov/help/means-tested-benefits
- See also: Government Shutdown Clock — https://www.whitehouse.gov/government-shutdown-clock/
- Available data/document: Individual Participant Data Set: 014/BR/612 — https://virtualtribunalmonastery.vhx.tv/ — Regarding an individual means test, the Holistic Healthcare needs exceed the costs associated with the service. As a licensed referral, ordering, and nonclinical prescribing Holistic Medicine provider only, cost-effective pastoral counseling serve its purpose.
- Available data/document: Study Protocol — https://www.ncbi.nlm.nih.gov/myncbi/goddess%20zena.jones.1/bibliography/public/

DOCUMENTS (3):
  • Study Protocol (2026-01-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT06098755/Prot_004.pdf
  • Statistical Analysis Plan (2026-01-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT06098755/SAP_005.pdf
  • Informed Consent Form (2025-10-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT06098755/ICF_003.pdf